CLINICAL TRIAL: NCT02546388
Title: Somatostatin Receptor Imaging in Patients With Suspected Cardiac Sarcoidosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marcelo F. Di Carli, MD, FACC (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor-Investigator, Marcelo F. Di Carli, MD, FACC, Chief of Nuclear Medicine, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015P001421
Record Dates: First submitted 2015-09-09; First posted 2015-09-10 (Estimated); Results first posted 2020-03-25 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Sarcoidosis
MeSH Terms: conditions — Sarcoidosis | interventions — pentetreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Indium-111 Pentreotide (OctreoScan) (Experimental): Patients with biopsy-proven extra-cardiac sarcoidosis OR atypical findings on FDG PET and MRI without previous biopsy will be recruited to receive an injection of the FDA-approved radiotracer Indium-111 Pentreotide (OctreoScan). The imaging protocol will consist of imaging at 4 and 24 hours after OctreoScan injection.
  Interventions: Drug: Indium-111 Pentreotide
- Gallium-68 DOTATATE (Experimental): Patients with biopsy-proven extra-cardiac sarcoidosis OR atypical findings on FDG PET and MRI without previous biopsy will be recruited to receive an injection of the FDA-approved radiotracer Gallium-68 DOTATATE. The imaging protocol will consist of imaging 1 hour after injection for DOTATATE.
  Interventions: Drug: Gallium-68 DOTATATE

INTERVENTIONS:
Drug: Indium-111 Pentreotide
  Other Names: OctreoScan
  Arms: Indium-111 Pentreotide (OctreoScan)
Drug: Gallium-68 DOTATATE
  Arms: Gallium-68 DOTATATE

SUMMARY:
The purpose of this research study to find out if a drug called OctreoScan or DOTATATE can help doctors diagnose people with cardiac sarcoidosis better.

OctreoScan and DOTATATE are both approved by the U.S. Food and Drug Administration (FDA) to diagnose certain tumors.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 or older
* Documentation of biopsy-proven sarcoidosis OR patients with typical findings on FDG PET and MRI without previous biopsy
* Clinical suspicion of cardiac involvement defined as the presence of any of the following: high-degree A-V nodal block, complete bundle branch block, reduced left or right ventricular systolic function, any cardiac arrhythmia, and/or unexplained chest pain, dyspnea or syncope
* PET/CT imaging demonstrating abnormal myocardial FDG uptake consistent with active inflammatory myocardium.

Exclusion Criteria:

* Initiation of steroids or any other immunosuppressive medication(s) following the completion of FDG-PET, as these medications, in theory, may subsequently suppress OctreoScan or DOTATATE uptake in the heart.
* Patients with history of neuroendocrine tumors (specially insulinomas)
* Patients taking the medication Octreotide
* Patients on total parenteral nutrition (TPN)
* Women who are pregnant or breastfeeding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-10; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Gallium-68 DOTATATE: Patients with biopsy-proven extra-cardiac sarcoidosis OR atypical findings on FDG PET and MRI without previous biopsy will be recruited to receive an injection of the FDA-approved radiotracer Gallium-68 DOTATATE. The imaging protocol will consist of imaging at 1 hour after injection for DOTATATE.
Period: Overall Study
Arm/Group | Indium-111 Pentreotide (OctreoScan) | Gallium-68 DOTATATE
Started | 4 | 13
Completed | 4 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indium-111 Pentreotide (OctreoScan) | Gallium-68 DOTATATE | Total
Number analyzed (Participants) | 4 | 13 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 8 | 11
  >=65 years | 1 | 5 | 6
Age, Continuous [Mean (Full Range); unit: Years] | 62 [54 to 73] | 59 [43 to 76] | 60 [43 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 1 | 11 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 13 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 3 | 13 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 13 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Characterized by Abnormal or Negative Uptake
Description: To correlate localization and number of increased radiotracer foci between FDG-PET and DOTATATE studies.
Time Frame: 1 hour
Population: We initially planned to do OctreoScan, but Dotatate became FDA approved in the process. Due to the superior image quality, lower radiation, and shorter protocol for Dotatate, we decided to abandon OctreoScan.
Measure: Count of Participants; unit: Participants
Arm/Group | Gallium-68 DOTATATE | Indium-111 Pentreotide (OctreoScan)
Number analyzed (Participants) | 13 | 0
Participants
  Number of Subjects with Definitely Abnormal Uptake | 4 |
  Number of Subjects with Probably Abnormal Uptake | 3 |
  Number of Subjects with Negative Uptake | 6 |

2. Secondary Outcome: Effect of Treatment
Description: To correlate localization and number of increased radiotracer foci between FDG-PET and DOTATATE studies.
Time Frame: 1 hour
Population: Only one patient underwent a repeat Dotatate PET/CT scan to investigate treatment response in our study
Measure: Count of Participants; unit: Participants
Groups:
- Participants With a Positive or Negative Response to Treatment: Patients with biopsy-proven extra-cardiac sarcoidosis OR atypical findings on FDG PET and MRI without previous biopsy will be recruited to receive an injection of the FDA-approved radiotracer Indium-111 Pentreotide (OctreoScan) or Gallium-68 DOTATATE. The imaging protocol will consist of imaging at 1 hour after injection for DOTATATE.
Arm/Group | Participants With a Positive or Negative Response to Treatment
Number analyzed (Participants) | 1
Participants
  Number of Subjects wPositive Response to Treatment | 1
  Number of Subjects wNegative Response to Treatment | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected until up to 4 days after the last visit. One subject completed the optional Study Day 2 visit, so adverse events were collected up to 6 months after consent.
Groups:
- Gallium-68 DOTATATE: Patients with biopsy-proven extra-cardiac sarcoidosis OR atypical findings on FDG PET and MRI without previous biopsy will be recruited to receive an injection of the FDA-approved radiotracer or Gallium-68 DOTATATE. The imaging protocol will consist of imaging at 1 hour after injection for DOTATATE.
Arm/Group | Indium-111 Pentreotide (OctreoScan) | Gallium-68 DOTATATE
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/13
Other Adverse Events (participants affected / at risk) | 0/4 | 0/13

LIMITATIONS AND CAVEATS:
Limitations include small sample size (we only included individuals with myocardial FDG uptake) and there is no gold standard for the diagnosis of inflammation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-13): https://cdn.clinicaltrials.gov/large-docs/88/NCT02546388/Prot_SAP_000.pdf